CLINICAL TRIAL: NCT00154102
Title: Open, Randomized, Controlled, Multicenter Phase III Study Comparing 5FU/ FA Plus Irinotecan Plus Cetuximab Versus 5FU/FA Plus Irinotecan as First-line Treatment for Epidermal Growth Factor Receptor-expressing Metastatic Colorectal Cancer
Brief Title: Cetuximab Combined With Irinotecan in First-line Therapy for Metastatic Colorectal Cancer (CRYSTAL)
Acronym: CRYSTAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Monika Foerster, Merck Serono
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-013
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Epidermal Growth Factor Receptor (EGFR) Expressing Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; EGFR; Irinotecan; cetuximab; first-line treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab Plus FOLFIRI (Experimental)
  Interventions: Drug: Cetuximab; Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan)
- FOLFIRI Alone (Active Comparator)
  Interventions: Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan)

INTERVENTIONS:
Drug: Cetuximab — Cetuximab intravenous infusion of 400mg/m^2 for the first infusion then weekly intravenous infusion of 250mg/m^2. Number of Cycles: until progression or unacceptable toxicity develops
  Arms: Cetuximab Plus FOLFIRI
Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan) — Bi-weekly Irinotecan infusion of 180mg/m^2, Folinic Acid infusion of 400mg/m^2 (racemic) or 200mg/m^2 (L-form), 5-Fluorouracil bolus of 400mg/m^2 followed by a 46-hour continuous infusion of 2400mg/m^2 Number of Cycles: until progression or unacceptable toxicity develops

SUMMARY:
Drugs used against cancer work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Giving combination chemotherapy together with cetuximab as first treatment after diagnosis of a metastatic colorectal cancer ('1st-line' treatment) may improve the treatment efficacy. However, it is not yet known whether giving combination chemotherapy together with cetuximab is more effective than combination chemotherapy alone. This open-label trial investigates the effectiveness of cetuximab in combination with a standard and effective chemotherapy (5-Fluorouracil (5FU)/Folinic acid (FA) plus irinotecan) for metastatic colorectal cancer in first-line setting, compared to the same chemotherapy alone on patient expressing the epidermal growth factor (EGF) receptor.

Patients expressing this EGF Receptor will be randomly assign in one of the 2 groups to either receive the combination chemotherapy alone or with cetuximab (open-label study) and will then be treated until progression of the disease or unacceptable toxicity occur. Regular efficacy assessments (every 8 weeks) based on imaging will be performed throughout the study together with regular safety assessments (e.g. safety labs). An independent Safety Board of experts will also monitor safety data.

After participant discontinuation from the trial, regular updates on further treatments and survival status will be requested from the investigator.

The entire study (from the first patient entering the study to the last collect of follow-up information) is 4-5 years long.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* Inoperable metastatic disease
* Immunohistochemical evidence of epidermal growth factor receptor expression in tumor tissue
* Presence of at least 1 bi-dimensionally measurable index lesion

Exclusion Criteria:

* Previous irinotecan-based chemotherapy
* Previous chemotherapy for colorectal cancer except adjuvant treatment if terminated more than 6 months before the start of study treatment
* Radiotherapy, surgery (excluding prior diagnostic biopsy) or any investigational drug in the 30 days before the start of study treatment
* Brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1221 (Actual)
Dates: Start 2004-05; Primary Completion 2006-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric van Cutsem, Professor, Principal Investigator — University Hospital Gasthuisberg, Department Internal Medicine, Leuven, Belgium
Locations (154):
- Research Site, Buenos Aires, Argentina
- Australia (6):
  - Research Site, Bedford Park
  - Research Site, Darlinghurst
  - Research Site, Heidelberg
  - Research Site, Nedlands
  - Research Site, West Perth
  - Research Site, Woodville
- Austria (8):
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Kufstein
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Sankt Veit an der Glan
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (7):
  - Research Site, Antwerp
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (4):
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovidiv
  - Research Site, Sofia
  - Research Site, Varna
- Chile (2):
  - Research Site, Santiago-Las Condes
  - Research Site, Santiago-Providencia
- Czechia (2):
  - Research Site, Chomutov
  - Research Site, Prague
- Research Site, Turku, Finland
- France (14):
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Colmar
  - Research Site, Grenoble
  - Research Site, La Roche-sur-Yon
  - Research Site, Lorient
  - Research Site, Marseille
  - Research Sites, Nantes
  - Research Site, Périgueux
  - Research Site, Rennes
  - Research Site, Saint-Grégoire
  - Research Site, Strasbourg
  - Research Site, Toulon
  - Research Site, Villejuif
- Germany (17):
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Homburg/Saar
  - Research Site, Jena
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Oldenburg
  - Research Site, Ulm
- Greece (3):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
- Hong Kong (2):
  - Research Site, Pokfulam
  - Research Site, Shatin
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Pécs
- Italy (12):
  - Research Site, Ancona
  - Research Site, Aviano
  - Research Site, Bari
  - Research Site, Benevento
  - Research Site, Florence
  - Research Site, Mantova
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
- Research Site, México, Mexico
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Apeldoom
  - Research Site, Blaricum
  - Research Site, Roosendaal
  - Research Site, The Hague
  - Research Site, Zwolle
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gliwice
  - Research Site, Krakow
  - Research Site, Opole
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (3):
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Suceava
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Research Site, Singapore, Singapore
- Slovakia (5):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Trnava
  - Research Site, Žilina
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Madrid
  - Research Site, Palma de Mallorca
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Chiayi City
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (9):
  - Research Site, Charkassy
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kiev
  - Research Site, Kryvyi Rih
  - Research Site, Luhansk
  - Research Site, Lviv
  - Research Site, Uzhhorod
  - Research Site, Zhaporozhye
- United Kingdom (10):
  - Research Site, Brighton
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, Kent
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Peterborough
  - Research Site, Rhyl
  - Research Site, Sutton

REFERENCES:
- [Result] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720
- [Result] Van Cutsem E, Lang I, Folprecht G, Nowacki M, Cascinu S, Shchepotin I, Maurel J, Cunningham D, Celik I, Kohne C Cetuximab plus FOLFIRI in the treatment of metastatic colorectal cancer (mCRC): The influence of KRAS and BRAF biomarkers on outcome: Updated data from the CRYSTAL trial. ASCO 2010 Gastrointestinal Cancers Symposium, Orlando, USA January 2010 Abstract No: 281
- [Result] Lang I, Kohne CH, Folprecht G, Nowacki MP, Cascinu S, Shchepotin I, Maurel J, Cunningham D, Zubel A, Van Cutsem E Cetuximab plus FOLFIRI in 1st-line treatment of metastatic colorectal cancer: Quality of life (QoL) analysis of patients (pts) with KRAS wild-type (wt) tumours in the CRYSTAL trial. European Journal of Cancer Supplements. 2009 7(2):345
- [Derived] Dercle L, Lu L, Lichtenstein P, Yang H, Wang D, Zhu J, Wu F, Piessevaux H, Schwartz LH, Zhao B. Impact of Variability in Portal Venous Phase Acquisition Timing in Tumor Density Measurement and Treatment Response Assessment: Metastatic Colorectal Cancer as a Paradigm. JCO Clin Cancer Inform. 2017 Nov;1:1-8. doi: 10.1200/CCI.17.00108. PMID 30657405
- [Derived] Tejpar S, Stintzing S, Ciardiello F, Tabernero J, Van Cutsem E, Beier F, Esser R, Lenz HJ, Heinemann V. Prognostic and Predictive Relevance of Primary Tumor Location in Patients With RAS Wild-Type Metastatic Colorectal Cancer: Retrospective Analyses of the CRYSTAL and FIRE-3 Trials. JAMA Oncol. 2017 Feb 1;3(2):194-201. doi: 10.1001/jamaoncol.2016.3797. PMID 27722750
- [Derived] Licitra L, Storkel S, Kerr KM, Van Cutsem E, Pirker R, Hirsch FR, Vermorken JB, von Heydebreck A, Esser R, Celik I, Ciardiello F. Predictive value of epidermal growth factor receptor expression for first-line chemotherapy plus cetuximab in patients with head and neck and colorectal cancer: analysis of data from the EXTREME and CRYSTAL studies. Eur J Cancer. 2013 Apr;49(6):1161-8. doi: 10.1016/j.ejca.2012.11.018. Epub 2012 Dec 19. PMID 23265711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject in: 10 Aug 2004/4 Nov 2005. Clinical cut-off efficacy analyses except survival: 27 Jul 2006, Cut off date IRC data: 14 Dec 2006; cut-off safety analyses: 30 Nov 2007; cut-off survival analyses: 31 May 2009; cut-off KRAS analyses: 28 Aug 2009.
  1221 subjects were randomised or treated, of whom 1198 were randomised and treated.
Pre-assignment Details: At the prescreening visit the subject completed the first informed consent form, and a sample of tumor tissue for determination of EGFR expression was to be obtained.
  The screening (baseline) visit was performed no more than 21 days before randomization. EGFR-expressing subjects completed a second informed consent form to participate in the study.
Groups:
- Cetuximab Plus FOLFIRI: Cetuximab intravenous infusion of 400mg/m^2 for the first infusion then weekly intravenous infusion of 250mg/m^2. Bi-weekly Irinotecan infusion of 180mg/m^2, Folinic Acid infusion of 400mg/m^2 (racemic) or 200mg/m^2 (L-form), 5-Fluorouracil bolus of 400mg/m^2 followed by a 46-hour continuous infusion of 2400mg/m^2 Number of Cycles: until progression or unacceptable toxicity develops
- FOLFIRI Alone: Bi-weekly Irinotecan infusion of 180mg/m^2, Folinic Acid infusion of 400mg/m^2 (racemic) or 200mg/m^2 (L-form), 5-Fluorouracil bolus of 400mg/m^2 followed by a 46-hour continuous infusion of 2400mg/m^2 Number of Cycles: until progression or unacceptable toxicity develops
Period: Overall Study
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Started | 599 (Randomized and treated subjects; 1 additional subject was treated but not randomised) | 599 (Randomized and treated subjects; 3 additional subjects were treated but not randomised)
Completed | 592 | 597
Not Completed | 7 | 2
Not completed — investigational study phase ongoing | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone | Total
Number analyzed (Participants) | 599 | 599 | 1198
Age, Continuous [Mean (Standard Deviation); unit: years] — Age missing for 1 subject
  years | 60.0 (10.52) | 59.8 (11.06) | 59.9 (10.79)
Age, Customized [Number; unit: participants] — Age missing for 1 subject
  participants
    Missing | 1 | 0 | 1
    Between 18 and 65 years | 374 | 377 | 751
    >=65 years | 224 | 222 | 446
Gender [Count of Participants; unit: Participants]
  Female | 230 | 243 | 473
  Male | 369 | 356 | 725
Region of Enrollment [Number; unit: participants]
  Western Europe | 262 | 267 | 529
  Eastern Europe | 203 | 201 | 404
  Rest of the World | 134 | 131 | 265

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Time - Independent Review Committee (IRC) Assessments
Description: Duration from randomization until radiological progression (based on modified World Health Organisation (WHO) criteria) or death due to any cause.
  Only deaths within 60 days of last tumor assessment are considered. Patients without event are censored on the date of last tumor assessment.
Time Frame: Time from randomisation to disease progression, death or last tumour assessment, reported between day of first patient randomised, 10 Aug 2004, until cut-off date, 27 July 2006
Population: Primary analysis on Intent to Treat (ITT) population i.e. all randomized subjects who have received at least one dose of randomized treatment (allocation to treatment groups as randomized).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 599 | 599
months | 8.9 [8.0 to 9.4] | 8.0 [7.6 to 9.0]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; The study was planned with 633 progression events, in order to provide 80% power to test the null hypothesis of no difference in PFS time between treatment groups, assuming a hazard ratio (HR) of 0.8 of cetuximab + chemotherapy (CTX) over CTX alone. Significance level was fixed at 5%. The two-sided stratified log-rank test was employed, considering the randomization strata (region: Western Europe, Eastern Europe, outside Europe and Karnovsky Performance Scale (KPS):<80 vs. ≥80); Test type: Superiority or Other; p = 0.0479, Stratified log rank; Kaplan-Meier method was used to estimate median PFS time. HR was calculated using Cox proportional hazards model stratified by randomization strata; Hazard Ratio (HR) = 0.853, 95% CI 2-sided [0.728 to 1.000]

2. Primary Outcome: Progression-free Survival Time (Chinese V-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Wild-Type Population) - Independent Review Committee (IRC) Assessments
Description: Duration from randomization until radiological progression (based on modified WHO criteria) or death due to any cause.
  Only deaths within 60 days of last tumor assessment are considered. Patients without event are censored on the date of last tumor assessment.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) population with KRAS Wild Type tumor status as collected until 28 August 2009
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 316 | 350
months | 9.9 [9.0 to 11.3] | 8.4 [7.4 to 9.2]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; The two-sided stratified log-rank test was employed at the 5% significance level, considering the randomization strata (region: Western Europe, Eastern Europe, outside Europe and KPS:<80 vs. ≥80); Test type: Superiority or Other; p = 0.0012, Stratified log rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.696, 95% CI 2-sided [0.558 to 0.867]

3. Primary Outcome: Progression-free Survival Time (KRAS Mutant Population) - Independent Review Committee (IRC) Assessments
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) population with KRAS Mutant tumor status as collected until 28 August 2009
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 214 | 183
months | 7.4 [6.1 to 8.0] | 7.7 [7.3 to 9.2]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2648, Stratified log rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.171, 95% CI 2-sided [0.887 to 1.544]

4. Secondary Outcome: Overall Survival Time (OS)
Description: Time from randomization to death. Patients without event are censored at the last date known to be alive or at the clinical cut-off date, whichever is later.
Time Frame: Time from randomisation to death or last day known to be alive, reported between day of first patient randomised, 10 Aug 2004, until cut-off date, 31 May 2009
Population: ITT population (allocation to treatment groups as randomized and treated)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 599 | 599
months | 19.9 [18.5 to 21.3] | 18.6 [16.7 to 19.8]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0419, Stratified log rank; Kaplan-Meier method was used to estimate median OS time. HR was calculated using Cox proportional hazards model stratified by randomization strata; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.774 to 0.995]

5. Secondary Outcome: Overall Survival Time (KRAS Wild-Type Population)
Description: as for outcome 4
Time Frame: Time from randomisation to death or last day known to be alive reported between day of first patient randomised, 10 Aug 2004, until cut-off date, 31 May 2009
Population: Intent to Treat (ITT) population with KRAS Wild Type tumor status as collected until 28 August 2009
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 316 | 350
months | 23.5 [21.2 to 26.3] | 20.0 [17.4 to 21.7]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0093, Stratified log rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.796, 95% CI 2-sided [0.670 to 0.946]

6. Secondary Outcome: Overall Survival Time (KRAS Mutant Population)
Description: as for outcome 4
Time Frame: as for outcome 5
Population: Intent to Treat (ITT) population with KRAS Mutant tumor status as collected until 28 August 2009
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 214 | 183
months | 16.2 [14.9 to 17.9] | 16.7 [14.9 to 19.4]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7549, Stratified log rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.035, 95% CI 2-sided [0.834 to 1.284]

7. Secondary Outcome: Best Overall Response Rate - Independent Review Committee (IRC) Assessments
Description: The best overall response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as the best overall response according to radiological assessments (based on modified WHO criteria).
Time Frame: evaluations were performed every 6 weeks until progression reported between day of first patient randomised, 10 Aug 2004, until cut-off date, 27 July 2006
Population: ITT population (allocation to treatment groups as randomized and treated)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 599 | 599
percentage of participants | 46.9 [42.9 to 51.0] | 38.7 [34.8 to 42.8]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; The two-sided stratified Cochran-Mantel-Haenszel (CMH) test was employed at the 5% significance level, considering the randomization strata (region: Western Europe, Eastern Europe, outside Europe and KPS:<80 vs. ≥80); Test type: Superiority or Other; p = 0.0038, Stratified cochran-mantel haenszel test; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.12 to 1.77]

8. Secondary Outcome: Best Overall Response Rate (KRAS Wild-Type Population) - Independent Review Committee (IRC) Assessments
Description: as for outcome 7
Time Frame: as for outcome 7
Population: Intent to Treat (ITT) population with KRAS Wild Type tumor status as collected until 28 August 2009
Measure: Number (95% Confidence Interval); unit: percentage participants
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 316 | 350
percentage participants | 57.3 [51.6 to 62.8] | 39.7 [34.6 to 45.1]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.069, 95% CI 2-sided [1.515 to 2.826]

9. Secondary Outcome: Best Overall Response Rate (KRAS Mutant Population) - Independent Review Committee (IRC) Assessments
Description: as for outcome 7
Time Frame: as for outcome 7
Population: Intent to Treat (ITT) population with KRAS Mutant tumor status as collected until 28 August 2009
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 214 | 183
percentage of participants | 31.3 [25.2 to 38.0] | 36.1 [29.1 to 43.5]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.3475, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.822, 95% CI 2-sided [0.544 to 1.242]

10. Secondary Outcome: Disease Control Rate - Independent Review Committee (IRC) Assessments
Description: The disease control rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease as best overall response according to radiological assessments (based on modified WHO criteria).
Time Frame: as for outcome 7
Population: ITT population (allocation to treatment groups as randomized and treated)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 599 | 599
percentage of participants | 84.3 [81.1 to 87.1] | 85.5 [82.4 to 88.2]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.6004, Stratified cochran-mantel haenszel test; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.67 to 1.26]

11. Secondary Outcome: Duration of Response - Independent Review Committee (IRC) Assessments
Description: Time from first assessment of Complete Response or Partial Response to disease progression or death (within 60 days of last tumor assessment).
  Patients without event are censored on the date of last tumor assessment. Tumor assessments based on modified WHO criteria.
Time Frame: Time from first assessment of complete response or partial response to disease progression, death or last tumor assessment reported between day of first patient randomised, 10 Aug 2004, until cut-off date, 27 July 2006
Population: ITT population (allocation to treatment groups as randomized and treated)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 599 | 599
months | 9.6 [9.1 to 12.9] | 7.7 [6.7 to 8.3]

12. Secondary Outcome: Participants With No Residual Tumor After Metastatic Surgery
Description: Participants with no residual tumor after on-study surgery for metastases
Time Frame: time from first dose up to 30 days after last dose of study treatment reported between day of first patient randomised, 10 Aug 2004, until cut-off date, 30 Nov 2007
Population: ITT population (allocation to treatment groups as randomized and treated)
Measure: Number; unit: Participants
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 599 | 599
Participants | 29 | 10
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFIRI vs FOLFIRI Alone; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.45 to 6.27]

13. Secondary Outcome: Quality of Life (QOL) Assessment European Organisation for the Research and Treatment of Cancer (EORTC) QLQ-C30 Global Health Status
Description: Mean global health status scores (EORTC QLQ-C30) against time for each treatment group. Scores were derived from mutually exclusive sets of items, with scale scores ranging from 0 to 100 after a linear transformation. Higher scores indicate a better QoL.
Time Frame: at baseline, at week 8, at week 16, at week 24, at week 32, and at week 40, reported between day of first patient randomised, 10 Aug 2004, until cut-off date, 27 July 2006
Population: 1125 subjects (566 Cetuximab + FOLFIRI; 559 FOLFIRI alone) completed at least 1 evaluable questionnaire & were included in the Evaluable for QLQ-C30 population. Numbers at each timepoint were (Cetuximab + FOLFORI/FOLFORI alone, respectively): baseline 430/423; Week 8 421/390; Week 16 312/309; Week 24 255/244; Week 32 164/154; Week 40 122/96
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 566 | 559
scores on a scale
  At baseline | 58.88 (1.185) | 60.33 (1.155)
  At week 8 | 59.02 (1.187) | 61.83 (1.176)
  At week 16 | 60.77 (1.276) | 63.29 (1.249)
  At week 24 | 61.83 (1.368) | 64.06 (1.364)
  At week 32 | 59.68 (1.590) | 65.07 (1.612)
  At week 40 | 63.43 (1.835) | 64.02 (1.991)

14. Secondary Outcome: Quality of Life Assessment (EORTC QLQ-C30) Social Functioning
Description: Mean social functioning scores (EORTC QLQ-C30) against time for each treatment group. Scores were derived from mutually exclusive sets of items, with scale scores ranging from 0 to 100 after a linear transformation. Higher scores indicate a higher level of functioning.
Time Frame: as for outcome 13
Population: 1125 subjects (566 in the Cetuximab + FOLFIRI arm and 559 in the FOLFIRI alone arm) completed at least one evaluable QLQ-C30 questionnaire and were thus included in the Evaluable for QLQ-C30 population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 566 | 559
scores on a scale
  At baseline | 75.21 (1.426) | 77.28 (1.395)
  At week 8 | 74.14 (1.430) | 76.71 (1.415)
  At week 16 | 73.72 (1.533) | 76.67 (1.498)
  At week 24 | 76.31 (1.644) | 77.98 (1.633)
  At week 32 | 74.04 (1.903) | 75.64 (1.933)
  At week 40 | 76.58 (2.198) | 78.07 (2.388)

15. Secondary Outcome: Safety - Number of Patients Experiencing Any Adverse Event
Description: Please refer to Adverse Events section for further details
Time Frame: as for outcome 12
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 600 | 602
participants | 599 | 597

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after the last dose of study treatment.
Description: Treatment-emergent adverse events were defined as those with onset occurring at or after the first dosing day of study medication and up to 30 days after the last administration of any study drug or the clinical cut-off date.
Groups:
- Cetuximab Plus FOLFIRI: Cetuximab intravenous infusion of 400mg/m^2 for the first infusion then weekly intravenous infusion of 250mg/m^2. Bi-weekly Irinotecan infusion of 180mg/m^2, Folinic Acid infusion of 400mg/m^2 (racemic) or 200mg/m^2 (L-form), 5-Fluorouracil bolus of 400mg/m^2 followed by a 46-hour continuous infusion of 2400mg/m^2 Number of Cycles: until progression or unacceptable toxicity develops.
  Safety population: includes all treated subjects.
- FOLFIRI Alone: Bi-weekly Irinotecan infusion of 180mg/m^2, Folinic Acid infusion of 400mg/m^2 (racemic) or 200mg/m^2 (L-form), 5-Fluorouracil bolus of 400mg/m^2 followed by a 46-hour continuous infusion of 2400mg/m^2 Number of Cycles: until progression or unacceptable toxicity develops.
  Safety population: includes all treated subjects
Arm/Group | Cetuximab Plus FOLFIRI | FOLFIRI Alone
Serious Adverse Events (participants affected / at risk) | 263/600 | 204/602
Other Adverse Events (participants affected / at risk) | 593/600 | 591/602
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus FOLFIRI (N=600) | FOLFIRI Alone (N=602)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 8
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 16 | 13
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 7
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 37 | 35
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2
PLATELET TOXICITY (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 0
ANGINA PECTORIS (Cardiac disorders) | 2 | 0
ARRHYTHMIA (Cardiac disorders) | 1 | 0
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 | 1
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 2
CARDIAC ARREST (Cardiac disorders) | 3 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 0
CONDUCTION DISORDER (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 3 | 1
PALPITATIONS (Cardiac disorders) | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
DIABETES INSIPIDUS (Endocrine disorders) | 1 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 | 13
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 2
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 | 1
ANAL FISTULA (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 3
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 6 | 2
DIARRHOEA (Gastrointestinal disorders) | 36 | 21
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
GASTRO-INTESTINAL FISTULA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 2
GASTROINTESTINAL HYPOMOTILITY (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 2 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 2 | 0
ILEUS (Gastrointestinal disorders) | 10 | 7
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 7 | 8
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 8 | 5
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PERITONEAL EFFUSION (Gastrointestinal disorders) | 0 | 1
PERITONITIS (Gastrointestinal disorders) | 0 | 2
PROCTALGIA (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 4
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 2
STOMATITIS (Gastrointestinal disorders) | 0 | 1
SUBILEUS (Gastrointestinal disorders) | 2 | 8
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 15 | 16
ASTHENIA (General disorders) | 6 | 5
CATHETER RELATED COMPLICATION (General disorders) | 1 | 2
CATHETER SITE HAEMATOMA (General disorders) | 0 | 1
CATHETER SITE INFLAMMATION (General disorders) | 2 | 0
CATHETER SITE PAIN (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 3 | 2
CHILLS (General disorders) | 5 | 2
DEATH (General disorders) | 2 | 0
DISEASE PROGRESSION (General disorders) | 1 | 0
EXTRAVASATION (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 8
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 | 1
INFLAMMATION (General disorders) | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1
INFUSION SITE EXTRAVASATION (General disorders) | 0 | 1
INFUSION SITE PAIN (General disorders) | 0 | 1
LOCALISED OEDEMA (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 3 | 2
PYREXIA (General disorders) | 26 | 21
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 | 0
BILIARY FISTULA (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1
DILATATION INTRAHEPATIC DUCT ACQUIRED (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 2
ANAPHYLACTIC REACTION (Immune system disorders) | 3 | 0
HYPERSENSITIVITY (Immune system disorders) | 4 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0
ABDOMINAL INFECTION (Infections and infestations) | 1 | 0
ABSCESS (Infections and infestations) | 1 | 0
ABSCESS INTESTINAL (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1
CATHETER RELATED INFECTION (Infections and infestations) | 8 | 1
CATHETER SEPSIS (Infections and infestations) | 3 | 0
CATHETER SITE INFECTION (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 3 | 0
CENTRAL LINE INFECTION (Infections and infestations) | 10 | 4
ERYSIPELAS (Infections and infestations) | 1 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 4 | 1
LISTERIOSIS (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 3
LUNG ABSCESS (Infections and infestations) | 0 | 1
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 1 | 2
OTITIS MEDIA CHRONIC (Infections and infestations) | 1 | 0
PELVIC ABSCESS (Infections and infestations) | 0 | 1
PERIANAL ABSCESS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 9 | 7
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 | 0
POSTOPERATIVE INFECTION (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
RETROPERITONEAL ABSCESS (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 4 | 1
SEPTIC SHOCK (Infections and infestations) | 3 | 0
SINUSITIS (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0
URINARY TRACT INFECTION (Infections and infestations) | 4 | 3
VARICELLA (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 1 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 | 1
INTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 | 2
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
STENT OCCLUSION (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 2 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 0 | 1
LABORATORY TEST ABNORMAL (Investigations) | 1 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 1
PLATELET COUNT DECREASED (Investigations) | 1 | 0
URINE ANALYSIS ABNORMAL (Investigations) | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 1
ANOREXIA (Metabolism and nutrition disorders) | 4 | 4
CACHEXIA (Metabolism and nutrition disorders) | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 16 | 12
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 2
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 13 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 | 0
ORAL INTAKE REDUCED (Metabolism and nutrition disorders) | 2 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
OVARIAN LOW MALIGNANT POTENTIAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 2 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
COMA (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 1 | 0
COORDINATION ABNORMAL (Nervous system disorders) | 0 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 2 | 0
EPILEPSY (Nervous system disorders) | 1 | 1
HEADACHE (Nervous system disorders) | 1 | 0
HEMIPARESIS (Nervous system disorders) | 2 | 0
LETHARGY (Nervous system disorders) | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 2 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 2 | 2
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 | 1
ACUTE CARDIO-VASCULAR INSUFFICIENCY (Cardiac disorders) | 0 | 1 — An organ system was assigned to this adverse event as required for posting on Clinicaltrials.gov - the organ system was not assigned in the Clinical Study Report
ACUTE GASTROENTERITIS (Infections and infestations) | 0 | 1 — An organ system was assigned to this adverse event as required for posting on Clinicaltrials.gov - the organ system was not assigned in the Clinical Study Report
ACUTE PNEUMONIA (Infections and infestations) | 1 | 0 — An organ system was assigned to this adverse event as required for posting on Clinicaltrials.gov - the organ system was not assigned in the Clinical Study Report
CIRCULATORY INSUFFICIENCY (Cardiac disorders) | 1 | 0 — An organ system was assigned to this adverse event as required for posting on Clinicaltrials.gov - the organ system was not assigned in the Clinical Study Report
INFECTION OF OSTEOSYNTHESIS IN RIGHT ANCLE (Infections and infestations) | 1 | 0 — An organ system was assigned to this adverse event as required for posting on Clinicaltrials.gov - the organ system was not assigned in the Clinical Study Report
THROMBUS//CLOT IN VEIN OF LEFT HAND CAUSING INFECTION (General disorders) | 1 | 0 — An organ system was assigned to this adverse event as required for posting on Clinicaltrials.gov - the organ system was not assigned in the Clinical Study Report
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 2
EUPHORIC MOOD (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 2 | 0
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 2 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 1
URETERIC OBSTRUCTION (Renal and urinary disorders) | 2 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
VAGINAL HAEMORRHAGE (Renal and urinary disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 4
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 20 | 10
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 1
ACNE (Skin and subcutaneous tissue disorders) | 2 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
CATARACT OPERATION (Surgical and medical procedures) | 1 | 0
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 1 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 9 | 5
EMBOLISM (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 5 | 3
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 1
ISCHAEMIA (Vascular disorders) | 0 | 1
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 1
PERIPHERAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
PHLEBITIS (Vascular disorders) | 0 | 1
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 4 | 4
VENA CAVA THROMBOSIS (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 2 | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus FOLFIRI (N=600) | FOLFIRI Alone (N=602)
NEUTROPENIA (Blood and lymphatic system disorders) | 272 | 249
LEUKOPENIA (Blood and lymphatic system disorders) | 127 | 120
ANAEMIA (Blood and lymphatic system disorders) | 121 | 127
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 31 | 20
LYMPHOPENIA (Blood and lymphatic system disorders) | 29 | 35
CONJUNCTIVITIS (Eye disorders) | 88 | 13
DIARRHOEA (Gastrointestinal disorders) | 377 | 353
NAUSEA (Gastrointestinal disorders) | 322 | 359
VOMITING (Gastrointestinal disorders) | 194 | 231
STOMATITIS (Gastrointestinal disorders) | 169 | 110
ABDOMINAL PAIN (Gastrointestinal disorders) | 142 | 154
CONSTIPATION (Gastrointestinal disorders) | 135 | 119
DYSPEPSIA (Gastrointestinal disorders) | 78 | 46
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 45 | 33
FATIGUE (General disorders) | 192 | 186
PYREXIA (General disorders) | 136 | 64
ASTHENIA (General disorders) | 110 | 112
MUCOSAL INFLAMMATION (General disorders) | 82 | 53
OEDEMA PERIPHERAL (General disorders) | 48 | 42
INJECTION SITE REACTION (General disorders) | 40 | 38
PARONYCHIA (Infections and infestations) | 107 | 3
NASOPHARYNGITIS (Infections and infestations) | 30 | 35
WEIGHT DECREASED (Investigations) | 94 | 52
ANOREXIA (Metabolism and nutrition disorders) | 169 | 149
HYPOKALAEMIA (Metabolism and nutrition disorders) | 58 | 30
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 42 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 38 | 55
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 30 | 23
HEADACHE (Nervous system disorders) | 64 | 55
DIZZINESS (Nervous system disorders) | 43 | 40
DYSGEUSIA (Nervous system disorders) | 41 | 45
INSOMNIA (Psychiatric disorders) | 57 | 53
COUGH (Respiratory, thoracic and mediastinal disorders) | 64 | 59
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 53 | 32
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 50 | 27
RASH (Skin and subcutaneous tissue disorders) | 270 | 23
ALOPECIA (Skin and subcutaneous tissue disorders) | 224 | 229
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 146 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 133 | 30
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 101 | 27
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 97 | 10
PRURITUS (Skin and subcutaneous tissue disorders) | 73 | 28
ACNE (Skin and subcutaneous tissue disorders) | 69 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 54 | 5
ERYTHEMA (Skin and subcutaneous tissue disorders) | 40 | 12
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 35 | 3
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 34 | 1
HYPERTENSION (Vascular disorders) | 46 | 36
PHLEBITIS (Vascular disorders) | 38 | 20
HYPOTENSION (Vascular disorders) | 32 | 20

LIMITATIONS AND CAVEATS:
A non-specific outcome measure 'Safety' was deleted from the entry in error. A replacement outcome was created. The outcome refers to adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other